CLINICAL TRIAL: NCT04828408
Title: Evaluation of Diaphragm Functions in Laparoscopic Bariatric Surgeries
Brief Title: Diaphragm Functions in Bariatric Surgeries
Status: Completed | Type: Observational
Sponsor: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Derya Karasu, MD, Assoc Prof., Turkiye Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 2019/02-16.derya
Record Dates: First submitted 2021-03-26; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Diaphragm Disease; Pulmonary Function Test; Ultrasonography; Bariatric Surgery; Anesthesia
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric surgery — Patients with a body mass index (BMI) ˃35, age interval of 18-65, and ASA score II-III undergoing laparoscopic bariatric surgery were included in the study. Patients with neuromuscular, cardiopulmonary, and cerebrovascular diseases, phrenic nerve damage or diaphragm paralysis, those who have undergone thoracic surgery, who could not communicate, who did not want to participate in the study, who used alcohol, those who needed postoperative intensive care, those who had surgical complications during surgery, and those who were switched to open surgery were not included in the study.

SUMMARY:
Obesity is an important public health problem all over the world, and its prevalence is increasing every year. In obesity, significant changes occur in the mechanical properties of the lungs and chest wall due to fat deposits in the mediastinum and abdominal cavities. Upper abdominal surgical procedures usually cause impairment of respiratory functions by affecting respiratory volume and capacity. The risk of postoperative pulmonary complications increases with the decrease in restrictive capacities, hypoxemia, and increased respiratory work. It may also be due to causes such as diaphragm dysfunction, postoperative pain, and surgical incision.Ultrasonography (USG) is a method accepted for evaluating the normal and pathological conditions of the diaphragm. M-mode is used to evaluate the anatomical and functional disorders of the diaphragm. The diaphragm evaluation is performed with the anterior approach in the supine position and with different respiratory maneuvers (sniffing, deep inspiration, normal inspiration).

The aim of the study was to evaluate the diaphragm function by using USG and spirometry methods in patients who underwent bariatric surgery and to investigate the effect of postoperative pain score on diaphragm function.

DETAILED DESCRIPTION:
Approval for this single-center, prospective, observational study was performed after the approval of the local Ethics Committee and informed consent from the patients.

Diaphragm ultrasonography was performed before general anesthesia, after general anesthesia in the recovery room, and at the postoperative 24th hour in normal breathing, deep inspiration, and sniffing position. For USG evaluation, while the patients sit in the supine position at an angle of 45⁰, the 2.5-7.5 Mhz convex probe is placed perpendicular to the intercostal spaces through the liver window on the anterior axillary line; The posterior part of the right hemidiaphragm was evaluated by directing it medially, cephalad and dorsally. Diaphragm movements in M-mode were evaluated after detection of the diaphragm in the B-mode. The inspiratory amplitude of the diaphragm (DIA: distance traveled by the diaphragm between the beginning and end of inspiration, cm) in M-mode, inspiratory velocity (IV= DIA/inspiratory time, cm/sec), and expiratory velocity (EV= DIA/expiratory time, cm/sec) measurements were made. VAS scores of the patients were questioned while performing USG.

Pulmonary function tests (PFT) of patients before surgery and the postoperative first day and FVC, FEV1, PEF, FEF25-75, and FEV1/FVC measurements have been recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a body mass index (BMI) ˃35,
* age interval of 18-65,
* ASA score II-III undergoing laparoscopic bariatric surgery

Exclusion Criteria:

* Patients with neuromuscular, cardiopulmonary, and cerebrovascular diseases,
* phrenic nerve damage or diaphragm paralysis,
* those who have undergone thoracic surgery,
* who could not communicate,
* who did not want to participate in the study,
* who used alcohol,
* those who needed postoperative intensive care,
* those who had surgical complications during surgery,
* those who were switched to open surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
diaphragm function | time from 10 minutes before anesthesia to 24 hours postoperatively
  change from baseline in diaphragm inspiratory amplitude at 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Yıldırım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No